CLINICAL TRIAL: NCT06641219
Title: Clinical Evaluation of Lutetium-177 Labeled BQ7876 for Targeting of Prostate-Specific Membrane Antigen
Brief Title: Clinical Evaluation of [177Lu]Lu-BQ7876 for Targeting of Prostate-Specific Membrane Antigen
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tomsk National Research Medical Center of the Russian Academy of Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: [177Lu]Lu-BQ7876
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Prostate Cancers
Keywords: Prostate-Specific Membrane Antigen; Prostate Cancers; [177Lu]Lu-BQ7876; Radioligand Therapy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: Open-label, exploratory, single centre study. The subjects will receive a single injection of the labeled tracer.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate cancer (Experimental): One single intravenous injection of [177Lu]Lu-BQ7876
  Interventions: Drug: One single intravenous injection of [177Lu]Lu-BQ7876

INTERVENTIONS:
Drug: One single intravenous injection of [177Lu]Lu-BQ7876 — One single intravenous injection of 600-800 MBq [177Lu]Lu-BQ7876 in prostate cancer patients.

SUMMARY:
The study should evaluate the biological distribution of [177Lu]Lu-BQ7876 in patients with prostate cancer.

The objective are:

1. To evaluate the content of [177Lu]Lu-BQ7876 in the blood of patients with prostate cancer at different time points after a single intravenous administration.
2. To assess the distribution of [177Lu]Lu-BQ7876 in normal tissues and tumors at different time points.
3. To evaluate dosimetry of [177Lu]Lu-BQ7876.
4. To study the safety and tolerability of the drug [177Lu]Lu-BQ7876 after a single injection.

DETAILED DESCRIPTION:
The overall goal is to study the effectiveness of prostate-specific membrane antigen targeting using Lutetium-177 - labeled BQ7876.

Phase I of the study:

Biodistribution, dosimetry, safety and tolerability of [177Lu]Lu-BQ7876 in patients with prostate cancer.

The main objectives of the study:

1. To evaluate the content of [177Lu]Lu-BQ7876 in the blood of patients with prostate cancer at different time points after a single intravenous administration.
2. To evaluate the distribution of [177Lu]Lu-BQ7876 in normal tissues and tumors in patients with prostate cancer at different time points after a single intravenous administration.
3. To evaluate dosimetry of [177Lu]Lu-BQ7876 based on the pharmacokinetic parameters of the drug after a single intravenous administration.
4. To study the safety of use and tolerability of the drug [177Lu]Lu-BQ7876 after a single intravenous administration in a diagnostic dosage.

Methodology:

Open-label, exploratory, single centre study. The subjects will receive a single injection of the labeled tracer.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 18 years of age
* Clinical and radiological diagnosis of prostate cancer with histological verification.
* White blood cell count: > 2.0 x 10^9/L
* Haemoglobin: > 80 g/L
* Platelets: > 50.0 x 10^9/L
* Bilirubin =< 2.0 times Upper Limit of Normal
* Serum creatinine: Within Normal Limits
* Blood glucose level not more than 5.9 mmol/L
* Subject is capable to undergo the diagnostic investigations to be performed in the study
* Informed consent

Exclusion Criteria:

* Active current autoimmune disease or history of autoimmune disease
* Active infection or history of severe infection within the previous 3 months (if clinically relevant at screening)
* Known HIV positive or chronically active hepatitis B or C
* Administration of other investigational medicinal product within 30 days of screening
* Ongoing toxicity > grade 2 from previous standard or investigational therapies, according to US National Cancer Institute's

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2024-10-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
[177Lu]Lu-BQ7876 blood сlearance | 48 hours
  Measurement of [177Lu]Lu-BQ7876 activity in patient blood samples at various time points: after 5, 10, 20, 40, 60 and 90 minutes, 2, 3, 24, 48 hours.
Gamma camera-based whole-body [177Lu]Lu-BQ7876 | 120 hours
  Whole-body [177Lu]Lu-BQ7876 uptake coinciding with normal organs and tissues will be assessed using gamma camera and calculated as percentage (%) of the injected dose of the radiopharmaceutical at 1, 4, 24, 48, 72, 120 hours after single injection.
SPECT/CT-based [177Lu]Lu-BQ7876 uptake in tumor lesions (SUVmean) | 120 hours
  [177Lu]Lu-BQ7876 uptake (SUVmean) with tumor lesions will be assessed using single-photon emission computed tomography and measured in SUVmean after 4, 48, 72 and 120 hours after single injection of radiopharmaceutical.

SECONDARY OUTCOMES:
Percent of cases with abnormal findings relative to baseline [Safety and Tolerability] | 48 hours
  The safety attributable to [177Lu]Lu-BQ7876 injections will be evaluated based on the assessments of physical examination, vital signs, and ECG (percent of cases with abnormal findings relative to baseline)
Percent of participants with abnormal laboratory values that are related to [177Lu]Lu-BQ7876 injection [Safety and Tolerability] | 48 hours
  The safety attributable to [177Lu]Lu-BQ7876 injections will be evaluated based on the blood and urine laboratory tests (percent of cases with abnormal findings relative to baseline)
Percent of participants with adverse events that are related to [177Lu]Lu-BQ7876 injection [Safety and Tolerability] | 48 hours
  The safety attributable to [177Lu]Lu-BQ7876 injections will be evaluated based on the rate of adverse events(percent of cases with abnormal findings relative to baseline)
Percent of participants requiring administration of medication due to side effects that are related to [177Lu]Lu-BQ7876 injection [Safety and Tolerability] | 48 hours
  The safety attributable to [177Lu]Lu-BQ7876 injections will be evaluated based on the rate of administration of concomitant medication (percent of cases with abnormal findings relative to baseline)

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir I Chernov, MD, Prof, Principal Investigator — Tomsk NRMC
Locations (1):
- TomskNRMC, Tomsk, Russia

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (text, tables, figures, and appendices), underlying the results of the trial, will be shared with researchers to achieve the aims in the approved proposal
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Proposals may be submitted up to 36 months following publication of the results of the trial. After 36 months, the data will be available in the Center's data ware house but without investigator support other than deposited metadata.
Access Criteria: Information regarding submitting proposals and accessing data may be requested from the principal investigator by e-mail.